CLINICAL TRIAL: NCT02386891
Title: Influence of Ambient Temperature on Food Intake Through a Randomized Control Trial in an Office Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: X140206006
Record Dates: First submitted 2015-03-06; First posted 2015-03-12 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Food Intake in 2 Thermal Environments
Keywords: food intake; indoor thermal environment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cold (Experimental): The cold treatment was 18-20°C (64.5-68°F), which is at the lower end of the thermalneutral zone in healthy adults.
  Interventions: Other: Thermal Environment
- Warm (Experimental): The warm treatment was 25-27°C (77-80.6°F), which is above the range of the thermalneutral zone.
  Interventions: Other: Thermal Environment

INTERVENTIONS:
Other: Thermal Environment

SUMMARY:
Based on preliminary data and previous studies, the investigators hypothesize that the ambient temperature experienced by an individual influences his or her food intake in males and females aged 19 to 30. Specifically, exposure to temperatures above the thermoneutral zone (TNZ) will decrease consumption in young adults in a sedentary situation. Researchers will execute a randomized control trial specifically testing thermal exposure and its effect on an individual's food consumption. Participants will receive and wear a t-shirt. They will have a thermal image taken of the inner canthus of their eye and middle finger nail bed, representing a baseline of core and peripheral temperatures, respectively. They will be randomized to either a colder environment (65°F) or a warmer environment (75°F) under the artifice of monitoring routine office work with abnormal temperature conditions. Their knowledge of the experiment will be limited until the end. They will experience this temperature while filling out paperwork and performing basic office tasks. After one hour, another thermal image will be taken. Each participant will be presented with a large, Mellow Mushroom cheese pizza and directed to eat at their leisure and subsequently finish the office tasks over the next hour. The participants will then be debriefed on the parameters of the experiment and body measurements will be taken at the end so as to prevent bias of the subject by limiting their food intake. The investigators will quantify energy intake by weighing remaining food and comparing to known caloric content by weight from bomb calorimetry tests. The infrared thermal images will determine whether the temperatures experienced were extreme enough to initiate a change in thermoregulation.

DETAILED DESCRIPTION:
Previous studies suggest increased time spent outdoors is associated with lower body mass index (BMI).1,2 . In addition, energy expenditure and hunger have been associated with exposure to heat or cold. Increased usage of central heating and air conditioning systems coupled with increased time spent indoors has created an environment where humans are expending less energy to regulate their body temperature.3 The human thermoneutral zone (TNZ) is the range of ambient temperatures in which a healthy adult can maintain body temperature without expending energy beyond the normal basal metabolic rate. Energy intake and expenditure are adjusted at temperatures above and below the TNZ.4 The temperature of the food, smell, time of consumption, and number of people present are established factors that influence food consumption in humans.5 In addition, evidence supports the role of the environment upon an individual's food intake. Wall color, lighting, and ambient noise, influence consumption preferences and quantities.6 Based on research in animal models, particularly mice and livestock,food intake and subsequently, weight gain is reduced in high ambient temperatures.7-10 In addition in young, physically active, healthy males, food intake is inversely proportional to TNZ.11 However, energy expenditure increases above and below the TNZ. These studies are based on extreme conditions, therefore there is a lack of information on how small changes in ambient temperature may affect food intake in the general human public. Recent research shows the effectiveness of small changes over time to lead to changes in consumption practices.12 Thus, altering the thermal environment subtly may lead to a greater understanding of long term effects in weight management. The investigators have previously examined the thermal environment of persons going about their daily lives in both urban and rural settings (X120217008). Preliminary analysis of the results suggest increased % body fat is associated with lower heat exposure.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  * Ages 19-35
  * Men and women

Exclusion Criteria:

* Exclusion Criteria:

  * Any food allergy, including, but not limited to lactose or gluten intolerance.
  * Religious affiliations that include specific food guidelines.
  * Personal dietary restrictions, including but not limited to veganism.
  * Participation in any weight-reduction program, weight-loss diet, or other special diet within the previous 3 months.
  * Weight loss or gain of >5% of body weight in the past 6 months for any reason except post-partum weight loss.
  * Currently taking medication that suppresses or stimulates appetite or that affects body weight, including oral anti-diabetic medications.
  * History of prior surgical procedure for weight control or liposuction.
  * Anyone currently taking statins.
  * Self report of high blood pressure (above 140 systolic, 90 diastolic)
  * Current smoker or quit smoking less than 6 months prior.
  * Any major disease, including:
  * Active cancer or cancer requiring treatment in the past 2 years (except nonmelanoma skin cancer).

    * Active or chronic infections, including self-reported HIV positivity and active tuberculosis.
    * Active cardiovascular disease or event including hospitalization or therapeutic procedures for treatment of heart disease (e.g., coronary artery bypass, percutaneous transluminal coronary angioplasty) in the past 6 months; New York Heart Association Functional Class >2 with respect to congestive heart failure; stroke or transient ischemic attack in the past 6 months.
    * Gastrointestinal disease, including self-reported chronic hepatitis or cirrhosis, any episode of alcoholic hepatitis or alcoholic pancreatitis within past year, inflammatory bowel disease requiring treatment in the past year, recent or significant abdominal surgery (e.g., gastrectomy).
    * Active renal disease.
    * Lung disease: chronic obstructive airway disease requiring use of oxygen.
    * Diagnosed diabetes (type 1 or 2).
    * Uncompensated or uncontrolled psychiatric disease (such as schizophrenia and bipolar disorder) that, in opinion of the investigators, would impede conduct of the trial or completion of procedures.
  * Self reported history of or current eating disorders
  * Conditions or behaviors likely to effect the conduct of the trial: unable or unwilling to give informed consent; unable to communicate with the pertinent staff; another household member is a participant or staff member in the trial; current or anticipated participation in another research project that would interfere with the offered session; unwilling to accept condition assignment by randomization
  * Currently taking antidepressant, steroid, or thyroid medication, unless dosage has been stable for at least 6 months.
  * Self-report of a recent or ongoing problem with drug abuse or addiction.
  * Self report of excessive alcohol intake, either acute or chronic, defined as any one of the following: 1) average consumption of 3 or more alcohol containing beverages daily; 2) consumption of 7 or more alcoholic beverages within a 24-hr period in the past 12 months
  * Pregnancy and childbearing: currently pregnant or less than 3 months post partum; currently nursing or within 6 weeks of having completed nursing; pregnancy anticipated during between time of screening and session date; unwilling to report possible or confirmed pregnancies promptly during the course of the trial;
  * Students in the Environmental Health Science Department, Nutrition Sciences School, Any student, trainee, or post-doctoral fellow who is directly or indirectly receiving funding from the Nutrition Obesity Research Center.
  * Any other conditions which, in opinion of the investigators, would adversely affect the conduct of the trial.

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Food intake (kcalories) | 1 hour
  Participants experienced the thermal environment for 1 hour and then were presented food (pizza) and had 1 hour to eat to their fill.

SECONDARY OUTCOMES:
Estimate of thermoregulation | 2 hours
  An infrared thermal camera took thermal images of partipants inner canthus and 3rd fingernail bed as estimates of core and peripheral temperature respectively. The difference between core minus peripheral temperature estimates whether heat dissipation has been initiated.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham School of Public Health, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Bernhard MC, Li P, Allison DB, Gohlke JM. Warm Ambient Temperature Decreases Food Intake in a Simulated Office Setting: A Pilot Randomized Controlled Trial. Front Nutr. 2015 Aug 24;2:20. doi: 10.3389/fnut.2015.00020. eCollection 2015. PMID 26322311